CLINICAL TRIAL: NCT05675436
Title: Observational Study Investigating the Mechanistic Effects of Mitapivat in Subjects With Sickle Cell Disease
Brief Title: Investigating the Mechanistic Effects of Mitapivat in Subjects With Sickle Cell Disease
Status: Active, not recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001061; 001061-H
Record Dates: First submitted 2023-01-06; First posted 2023-01-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-27

CONDITIONS: Sickle Cell Anemia; Sickle Cell Thalassemia; Sickle Cell Pain; Hbss; Hbsc; Sickle Beta Thalassemia; Sickle Beta Zero Thalassemia; Sickle Cell Syndrome Variant
Keywords: Sickle Cell Pain Crisis; Sickle Cell Anemia; Sickle Cell Treatment; Sickle Cell Therapy; Hemoglobin; Natural History
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: i. Phase 3: Mitapivat 50 mg BID
- 2: ii. Phase 3: Mitapivat 100 mg BID
- 3: iii. Phase 3: Mitapivat Open-Label Extension Period

SUMMARY:
Background:

Sickle cell disease (SCD) is an inherited blood disorder. The disease affects the ability of red blood cells to carry oxygen; this in turn can injure organs including the heart, lungs, and kidneys. SCD can lead to serious illness and death. Treatments such as bone marrow transplants and gene therapies can cure SCD, but they are not widely available. Current drug treatments for SCD are not always effective. This natural history study will examine how a study drug (mitapivat) affects red blood cells in people with SCD.

Objective:

To learn how mitapivat affects red blood cells in people with SCD.

Eligibility:

People with SCD who are enrolled in the parent study, NIH protocol IRB001565-H.

Design:

Procedures for this study will be done during visits already scheduled for the parent study.

Participants will have additional blood drawn during study visits. The additional amount will be about 3.5 teaspoons.

Participants will undergo a test called near infrared spectroscopy (NIRS) up to 9 times. Probes will be placed on their skin. A blood pressure cuff will be placed on their arm. The cuff will be filled with air for up to 5 minutes and then released. Participants may be asked to breathe at a certain rate or to hold their breath during these measurements. NIRS measures oxygen levels, blood flow, and the makeup of skin and muscle.

Researchers will draw additional information for this study from participants medical records.

DETAILED DESCRIPTION:
Study Description:

Subjects actively enrolled protocol AG348-C-020 (NIH protocol IRB001565-H), an industry-sponsored phase 2/3 study investigating the efficacy of mitapivat in treating sickle cell disease (SCD), will be invited to participate in this protocol simultaneously to further investigate the mechanistic effects of mitapivat. Subjects will be asked for a blood sample at study visits and undergo near infrared spectroscopy (NIRS) testing to investigate the mechanisms of action of mitapivat in subjects with SCD.

Objectives:

To evaluate the mechanisms of action of mitapivat in subjects with SCD.

Endpoints:

PRIMARY ENDPOINT DURING BLINDED PERIOD:

The percentage change in the oxygen affinity measure p50 (defined as the partial pressure of oxygen at which Hb is 50% saturated with oxygen) between baseline and the average value at 12, 24 and 52 weeks. This change will be compared between the placebo and mitapivat arms.

PRIMARY ENDPOINTS DURING OPEN LABEL EXTENSION (OLE):

* Evaluate the effect of mitapivat by comparing inter-patient and intra-patient changes between year one and year two.
* Evaluate the effects of long term use of mitapivat in patients who were randomized onto mitapivat during the first year of the study.
* Evaluate the intra-patient changes for patients who were randomized onto the placebo during the first year of the study and transition to mitapivat during year two.

SECONDARY ENDPOINTS DURING BLINDED PERIOD:

* The p50 changes will also be assessed at the individual time points of 12, 24, and 52 weeks.
* Percentage of sickled cells and time to 50% sickling (t50) under normal and hypoxic ex vivo conditions at regular time intervals on mitapivat and percentage change from baseline to the individual time points at 12, 24, and 52 weeks. This change will be compared between the placebo and mitapivat arms.
* Percentage change in intracellular reactive oxidative species (ROS) in red blood cells (RBCs) using a ROS sensitive fluorescent probe and mass spectrometry- based proteomics of RBC lysates between baseline and the individual time points at 12, 24, and 52 weeks. This change will be compared between the placebo and mitapivat arms.
* The percentage change in phosphatidylserine (PS) externalization using annexin V labeling (marker of red cell survival) by flow cytometry between baseline and the individual time points at 12, 24, and 52 weeks. This change will be compared between the placebo and mitapivat arms.
* Percentage change in muscle physiology, tissue oxygenation and blood flow using NIRS methodologies between baseline the individual time points at 12, 24, and 52 weeks. This change will be compared between the placebo and mitapivat arms.
* RBC deformability and sickling using osmotic and oxygen gradient ektacytometry

TERTIARY/EXPLORATORY ENDPOINTS DURING BLINDED PERIOD:

* Evaluate effect of mitapivat on RBC metabolomics and proteomics between baseline and various follow-up periods. This change will be compared between the placebo and mitapivat arms.
* Measurement of glycated Hb S level as a surrogate measure for red cell half-life between baseline and various follow-up periods. This change will be compared between the placebo and mitapivat arms.
* Evaluate effect of mitapivat on RBC band 3 tyrosine phosphorylation between baseline and various follow-up periods.

This change will be compared between the placebo and mitapivat arms.

* Correlation between potential exploratory biomarkers and clinical laboratory parameters.
* Evaluate change in cerebral hemodynamic measurements through magnetic resonance imaging (MRI) for cerebral blood flow, oxygen extraction fraction, and cerebral metabolic rate of oxygen consumption from baseline, at 12 and 52 weeks. This change will be compared between the placebo and mitapivat arms.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects enrolled at NIH meeting eligibility for the parent study (AG348-C-020) are eligible for this study.

EXCLUSION CRITERIA:

Subjects that did not meet eligibility criteria to the parent protocol (AG348-C-020) will not be eligible to enroll for this study.

Subjects will be screened for implanted metal objects or devices that may be incompatible with MRI (i.e. cerebral aneurysm clip, cochlear implant, pacemaker, etc.) These subjects will be eligible to proceed with study enrollment, but will not undergo the optional MRI study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2027-10-27 (Estimated); Study Completion 2027-10-27 (Estimated)

PRIMARY OUTCOMES:
The percentage change in the oxygen affinity measure p50 (defined as the partial pressure of oxygen at which Hb is 50% saturated with oxygen) between baseline. | 12, 24 and 52 weeks
  This change will be compared between the placebo and mitapivat arms.

SECONDARY OUTCOMES:
The percentage change in phosphatidylserine (PS) externalization using annexin V labeling (marker of red cell survival) by flow cytometry between baseline and the individual time points | 12, 24, and 52 weeks
  This change will be compared between the placebo and mitapivat arms.
The p50 changes will also be assessed at the individual time points | 12, 24, and 52 weeks
  This change will be compared between the placebo and mitapivat arms.
Percentage change in muscle physiology, tissue oxygenation and blood flow using NIRS methodologies between baseline the individual time points | 12, 24, 52, and 59 weeks
  This change will be compared between the placebo and mitapivat arms.
Percentage of sickled cells and time to 50% sickling (t50) under normal and hypoxic ex vivo conditions at regular time intervals on mitapivat and percentage change from baseline to the individual time points | 12, 24, and 52 weeks
  This change will be compared between the placebo and mitapivat arms.
Percentage change in intracellular reactive oxidative species (ROS) in red blood cells (RBCs) using a ROS sensitive fluorescent probe and mass spectrometry- based proteomics of RBC lysates between baseline and the individual time points | 12, 24, and 52 weeks
  This change will be compared between the placebo and mitapivat arms.
RBC deformability and sickling using osmotic and oxygen gradient ektacytometry | 12, 24, and 52 weeks
  This change will be compared between the placebo and mitapivat arms.

CONTACTS AND LOCATIONS:
Overall Officials: Swee Lay Thein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided: It is not yet known if there will be a plan to make IPD available

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001061-H.html